CLINICAL TRIAL: NCT00340886
Title: Environmental Polymorphism Study (EPS)
Brief Title: NIEHS/UNC Environmental Polymorphism Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902004; 02-E-N004
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-19

CONDITIONS: Genetic Polymorphisms
Keywords: Genetic Susceptibility; Single Nucleotide Polymorphism; Environmental Risk Factor; Allelic Variants; Ascertainment by Genotype
MeSH Terms: conditions — Genetic Predisposition to Disease

SUMMARY:
The Environmental Genome Project (EGP) has completely or partially resequenced the protein coding and regulatory regions of 53 environmentally sensitive genes from 72 anonymous individuals of varying ethnic backgrounds to date. Some of the same genes have been resequenced in an additional set of 20 samples, and, in a subset of these, the introns and promoter regions have been sequenced as well. Within this population, 523 allelic variants (genetic polymorphisms), mostly single nucleotide polymorphisms (SNPs), have been found to date. If the polymorphism alters the behavior or expression of the encoded protein, it might be of clinical significance.

The Office of Clinical Research is planning to establish a large resource bank of frozen DNA samples (20,000) and make it available to NIEHS intramural investigators involved in the EGP to screen for the presence of these SNPs and other mutations by standard genotyping methods. To investigate the feasibility of such a large collection of samples, we plan to first conduct a pilot study to estimate the accrual rate and uncover potential problems that may be encountered in the larger effort. This IRB proposal is for the pilot study in which we will collect whole blood samples (EDTA-anticoagulated) from 481 patients at UNC Medical Center. Once the pilot study is complete, we will decide whether to proceed with the larger, 20,000 sample collection and if so, develop and submit for review a new IRB protocol for its implementation taking date from the pilot study into account.

For both the pilot study and larger, 20,000 sample collection, only blood left over from patients already having their blood drawn for hematology (complete blood count or CBC) assays as part of their routine clinical management will be used, thus eliminating the need to collect extra blood. Once the samples have been obtained from the clinical hematology laboratory and processed, they will be identifiable only with a unique identification number and sent to an NIEHS contractor (BioServe Biotechnlolgies, Laurel, MD) for DNA isolation.

During recruitment, interviewers will explain the study to potential participants, obtain their signatures on the informed consent documents, and answer any questions they have concerning this study. At this time, potential participants will be informed that, depending on the results of the genetic analyses of their blood samples, they may be recontacted at a later date and asked to participate in follow-up genotype/phenotype studies. These follow-up studies will be separate from this protocol and the subjects of future IRB proposals. The ultimate objective of these sample collections, combined with the follow-up genotype/phenotype studies, is to identify groups of individuals with genetic polymorphisms in environmentally sensitive genes, and to correlate their genotype with their clinical phenotype, a process known as "ascertainment by genotype."

DETAILED DESCRIPTION:
The Environmental Genome Project (EGP) has completely or partially resequenced the protein coding and regulatory regions of 53 environmentally sensitive genes from 72 anonymous individuals of varying ethnic backgrounds to date. Some of the same genes have been resequenced in an additional set of 20 samples, and, in a subset of these, the introns and promoter regions have been sequenced as well. Within this population, 523 allelic variants (genetic polymorphisms), mostly single nucleotide polymorphisms (SNPs), have been found to date. If the polymorphism alters the behavior or expression of the encoded protein, it might be of clinical significance.

The Program in Clinical Research is planning to establish a large resource bank of frozen DNA samples (20,000) and make it available to NIEHS intramural investigators involved in the EGP to screen for the presence of these SNPs and other mutations by standard genotyping methods. To investigate the feasibility of such a large collection of samples,

we plan to first conduct a pilot study to estimate the accrual rate and uncover potential problems that may be encountered in the larger effort. This IRB proposal is for the pilot study in which we will collect whole blood samples (EDTA-anticoagulated) from 481 patients at UNC Medical Center. Once the pilot study is complete, we will decide whether to proceed with the larger, 20,000 sample collection and if so, develop and submit for review a new IRB protocol for its implementation taking data from the pilot study into account.

For both the pilot study and larger, 20,000 sample collection, only blood left over from patients already having their blood drawn for hematology (complete blood count or CBC) and hemoglobin A1c (HbA1c) assays as part of their routine clinical management will be used, thus eliminating the need to collect extra blood. Once the samples have been obtained from the clinical laboratory and processed, they will be identifiable only with a unique identification number and sent to an NIEHS contractor (BioServe Biotechnlolgies, Laurel, MD) for DNA isolation.

During recruitment, interviewers will explain the study to potential participants, obtain their signatures on the informed consent documents, and answer any questions they have concerning this study. At this time, potential participants will be informed that, depending on the results of the genetic analyses of their blood samples, they may be recontacted at a later date and asked to participate in follow-up genotype/phenotype studies. These follow-up studies will be separate from this protocol and the subjects of future IRB proposals. The ultimate objective of these sample collections, combined with the follow-up genotype/phenotype studies, is to identify groups of individuals with genetic polymorphisms in environmentally sensitive genes, and to correlate their genotype with their clinical phenotype, a process known as "ascertainment by genotype."

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be greater than or equal to 18 years of age and currently having their blood drawn for a CBC and/or a HbA1c assay.

There are no health status criteria for participating in this study; patients may be healthy or have preexisting conditions.

EXCLUSION CRITERIA:

Patients will not be excluded based on gender, ethnicity, race or religion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2001-10-01; Study Completion 2010-05-19

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina Medical Center, Chapel Hill, North Carolina, United States